CLINICAL TRIAL: NCT00561769
Title: Growth Hormone co-Treatment Within a GnRH Agonist Long Protocol in Patients With Poor Ovarian Response
Brief Title: Luteal Phase Commencing of Growth Hormone
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Collaborators: Ren-Tıp ART Center, Bursa, Turkey (Unknown)
Other Study IDs: GATA 2005-21
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Last update posted 2007-11-21 (Estimated); Status verified 2007-11

CONDITIONS: Infertility
Keywords: poor responder; growth hormone; luteal
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: poor responder
  Interventions: Drug: Norditropin pen

INTERVENTIONS:
Drug: Norditropin pen — 12 IU per day

SUMMARY:
Commencing of growth hormone in luteal phase when follicular cohort for the next cycle is being gathered may increase mature oocytes in poor responder

ELIGIBILITY:
Inclusion Criteria:

* Poor responder

Exclusion Criteria:

* FSH >20 IU

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: poor response to previous COH in the same center
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2005-01; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
mature oocyte number | 2 years

SECONDARY OUTCOMES:
pregnancy rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Kucuk, Assoc Prof, Study Director — GATA Ankara
Locations (1):
- Ren Tıp ART Center, Bursa, Turkey (Türkiye)